CLINICAL TRIAL: NCT04779736
Title: Mitigating Sexual Stigma Within Healthcare Interactions to Improve Engagement of MSM in HIV Prevention
Brief Title: Mitigating Sexual Stigma Within Healthcare Interactions Improve Engagement of MSM in HIV Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Columbia University (Other); New York State Psychiatric Institute (Other); GMR Transcription (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2023-14892; K23MH124569 (NIH)
Record Dates: First submitted 2021-01-21; First posted 2021-03-03 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Human Immunodeficiency Virus; Stigma, Social; Patient Engagement
Keywords: Implementation science; Health stigma and discrimination framework; Theoretical domains framework; Theory and techniques tool; Anal sex stigma; Men who have sex with men; Sexual and gender minority
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Social Stigma; Patient Participation; Homosexuality; Coitus

STUDY DESIGN:
Intervention Model Description: This is a single group study. Sequential explanatory mixed methods pre/post design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pre-post design (Other): The pilot intervention will be evaluated using a pre-post design.
  Interventions: Behavioral: A set of implementation strategies to reduce sexual stigma

INTERVENTIONS:
Behavioral: A set of implementation strategies to reduce sexual stigma — The set of implementation strategies was finalized based on formative interviews and consultation with an advisory board. This included an in-person workshop for skills development, environmental restructuring through a website of information resources for healthcare consumers and HCWs, and supportive coaching components (i.e., coaching calls, an optional email listserve) and quality improvement meetings with two clinics to encourage and respond to the implementation of recommended practices.

SUMMARY:
The purpose of this study is to explore drivers and mitigators of anal sex stigma in healthcare, and then to develop and pilot an intervention for health workers that mitigates the deterrent effects of this stigma on the engagement of gay and bisexual men in HIV-related services.

DETAILED DESCRIPTION:
This 5-year study aims to understand determinants that perpetuate and mitigate stigma toward anal sex during healthcare encounters, in order to develop and pilot a strategy that responds to these determinants and thereby improves the quality of care and HIV service engagement among men who have sex with men (MSM). The study team collected data during in-depth interviews with 20 adult MSM as well as 20 adult healthcare workers (HCWs) to identify strategies that could be readily used in health services to reduce stigma. Analysis of this data then informed consultation with an advisory board of HCWs and healthcare consumers (not limited to MSM), to develop the content of a set of implementation strategies to mitigate stigma and thereby improve health service delivery. Evaluation of a set of implementation strategies was performed in the Southern US, a high incidence region, by pilot testing with 65 adult HCWs who in clinical sites where MSM are under-engaged in HIV services.

ELIGIBILITY:
MSM Participants

Inclusion Criteria:

1. be aged 18 or older
2. report being assigned male at birth and identifying currently as male
3. reside in the United States
4. read and communicate in English
5. have had anal intercourse with a man in the past year or intend to in the next year Exclusion Criteria: Not applicable

Healthcare Worker Participants

Inclusion Criteria:

1. be aged 18 or older
2. read and communicate in English
3. bear a role responsibility for HIV-related screening and referral (e.g., as a peer/outreach worker, test counselor, case manager, social worker, medical assistant, nurse, physician assistant, physician) Exclusion Criteria: Not applicable

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — For the formative phase of in-depth interviews, we required MSM to identify as adult and male and to report being assigned male at birth. Formative in-depth interviews with healthcare workers, advisory board membership, and pilot evaluation required no specific gender eligibility requirements.
Enrollment: 113 (Actual)
Dates: Start 2021-08-23 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Acceptability, appropriateness, and feasibility of the website component as assessed by the AFAS | Post-intervention, 1 week after completion of all implementation strategies
  Quantitative assessment using the 13-item Acceptability, Feasibility, & Appropriateness Scale (AFAS), with three subscales for each construct. Acceptability refers to satisfaction with the implementation strategies. Feasibility refers to compatibility of recommended practices with participants' current practices. Appropriateness refers to perceived fit with participants' work mission and goals. Mean scores for individual items and mean scores for subscales will reflect the response category range from 1 (Not at all) to 5 (Extremely), with higher scores indicating, respectively, greater acceptability, appropriateness and feasibility.
Acceptability, appropriateness, and feasibility of the in-person skills development workshop as assessed by the AFAS | Post-intervention, 1 week after completion of the in-person workshop
  Quantitative assessment using the 13-item Acceptability, Feasibility, & Appropriateness Scale (AFAS), with three subscales for each construct. Acceptability refers to satisfaction with the implementation strategies. Feasibility refers to compatibility of recommended practices with participants' current practices. Appropriateness refers to perceived fit with participants' work mission and goals. Mean scores for individual items and mean scores for subscales will reflect the response category range from 1 (Not at all) to 5 (Extremely), with higher scores indicating, respectively, greater acceptability, appropriateness and feasibility.
Acceptability of the in-person skills development workshop as assessed by the AARP | Post-intervention, 1 week after completion of the in-person workshop
  Quantitative assessment using the 8-item Abbreviated Acceptability Rating Profile (AARP). Acceptability refers to satisfaction with the implementation strategies. Mean scores for individual items and mean scores for the overall scale will reflect the response category range from 0 (Strongly disagree) to 5 (Strongly agree), with higher scores indicating, respectively, greater acceptability.
Determinants of implementation of the in-person skills development workshop as assessed by the DIBQ | Post-intervention 1 week after completion of the in-person workshop
  Quantitative assessment using a 25-item adaptation to the Determinants of Implementation Behavior Questionnaire (DIBQ). The DIBQ measures multiple domains from within the Theoretical Domains Framework (e.g., behavioral control, reinforcement) that are posited as determinants of implementation. Mean scores for individual items and mean scores for subscales will reflect the response category range, from 1 (Very difficult) to 7 (Very easy), with higher scores indicating greater positive valence related to that domain.
Acceptability, appropriateness, and feasibility of the coaching calls as assessed by the AFAS | Post-intervention, 1 week after completion of all implementation strategies
  Quantitative assessment using the 13-item Acceptability, Feasibility, & Appropriateness Scale (AFAS), with three subscales for each construct. Acceptability refers to satisfaction with the implementation strategies. Feasibility refers to compatibility of recommended practices with participants' current practices. Appropriateness refers to perceived fit with participants' work mission and goals. Mean scores for individual items and mean scores for subscales will reflect the response category range from 1 (Not at all) to 5 (Extremely), with higher scores indicating, respectively, greater acceptability, appropriateness and feasibility.
Acceptability, appropriateness, and feasibility of the quality improvement meetings as assessed by the AFAS | Post-intervention, 1 week after completion of all implementation strategies
  Quantitative assessment using the 13-item Acceptability, Feasibility, & Appropriateness Scale (AFAS), with three subscales for each construct. Acceptability refers to satisfaction with the implementation strategies. Feasibility refers to compatibility of recommended practices with participants' current practices. Appropriateness refers to perceived fit with participants' work mission and goals. Mean scores for individual items and mean scores for subscales will reflect the response category range from 1 (Not at all) to 5 (Extremely), with higher scores indicating, respectively, greater acceptability, appropriateness and feasibility.
Acceptability, appropriateness, and feasibility of the set of implementation strategies as assessed by qualitative interviews | Post-workshop (1 week after delivery of the in-person workshop) and post-intervention ( 1 week after completion of all implementation strategies
  Acceptability, appropriateness, and feasibility will be assessed through in-depth interviews following completion of quantitative assessments, as part of an explanatory sequential mixed-methods design.
Changes to determinants of implementation behavior as assessed by the DIBQ | (1) Baseline, pre-intervention, (2) Post-intervention 1 week after completion of the in-person workshop, (3) Post-intervention 1 week after completion of all implementation strategies
  Quantitative assessment using a 26-item adaptation to the Determinants of Implementation Behavior Questionnaire (DIBQ). The DIBQ measures multiple domains from within the Theoretical Domains Framework (e.g., role responsibility, confidence, positive and negative emotions) that are posited as mechanisms of action that mediate behavior change among health care workers. Mean scores for individual items and mean scores for subscales will reflect the response category range, from 1 (Very difficult) to 7 (Very easy), with higher scores indicating ease related to that domain.
Changes to knowledge about anal health and sexuality as assessed by the iASK | (1) Baseline, pre-intervention, (2) Post-intervention 1 week after completion of the in-person workshop, (3) Post-intervention 1 week after completion of all implementation strategies
  Quantitative assessment using the 10-item Inventory of Anal Sex Knowledge (iASK). The iASK measures knowledge as a potential mediator of behavior change. All items are scored as True/False for a total percentage of correct responses, ranging from 0-10, with higher scores indicating greater knowledge.
Changes to self-efficacy offering social support as assessed by the MOS-SSS Informational and Emotional Social Support Subscale | (1) Baseline, pre-intervention, (2) Post-intervention 1 week after completion of the in-person workshop, (3) Post-intervention 1 week after completion of all implementation strategies
  Quantitative assessment using 8 items adapted from the Medical Outcomes Study Social Support Survey to measure changes in self-efficacy offering social support (e.g., Be someone to give information to help a client understand a situation involving anal sex). Mean scores for individual items will reflect the response category range, from 1 (Very easy) to 5 (Very difficult), with lower scores indicating greater self-efficacy offering informational and emotional social support.
Changes to comfort discussing anal health and sexuality as assessed by 10 study-specific items | (1) Baseline, pre-intervention, (2) Post-intervention 1 week after completion of the in-person workshop, (3) Post-intervention 1 week after completion of all implementation strategies
  Quantitative assessment using 10 items developed for the current study to measure changes to comfort discussing anal health and sexuality with clients (e.g., Asking clients about their sexual orientation; Asking clients about their anal sex practices; Initiating a conversation about anal health; Asking clients about their specific questions or concerns related to anal health). Mean scores for individual items will reflect the response category range, from 0 (Not at all comfortable) to 6 (Very comfortable), with higher scores indicating greater comfort related to that activity.
Changes to the quality of care as assessed by 10 study-specific items | (1) Baseline, pre-intervention, (2) Post-intervention 1 week after completion of all implementation strategies
  Quantitative assessment using 10 items developed for the current study to measure changes to frequency of discussing quality of care with clients (e.g., Asking clients about their sexual orientation; Asking clients about their anal sex practices; Initiating a conversation about anal health; Asking clients about their specific questions or concerns related to anal health). Mean scores for individual items will reflect the response category range, from 0 (Not at all comfortable) to 6 (Very comfortable), with higher scores indicating greater reported frequency of each activity.
Changes to the engagement in HIV-related services as measured by electronic health record (EHR) in two HIV service delivery sites | (1) the 3-month period pre-intervention, (2) the 3-month period during intervention, and then (3) the 3-month post-intervention, up to 9 months total.
  In two HIV service delivery sites, among all sites involved in the study, engagement of clients will be assessed via EHR by measuring the number over the past 30 days of patients who have sought (a) HIV testing, (b) screening for PrEP eligibility, (c) received anogenital cytology for sexually transmitted infection. EHR will also be reviewed to assess documentation of (a) anal health conditions, (b) sexual history and (c) sexual behavior.
Impact of implementation strategies on the quality of care and engagement of clients as assessed by qualitative interviews | Post-intervention 1 month after completion of all implementation strategies
  Impact of the implementation strategies (i.e., website and environmental restructuring, in-person workshop, coaching calls, email listserv, and any additional implementation strategies developed over the course of the study) assessed through in-depth interviews following completion of quantitative assessments, as part of an explanatory sequential mixed-methods design.

CONTACTS AND LOCATIONS:
Overall Officials: Bryan Kutner, PhD, MPH, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Albert Einstein College of Medicine, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2023-10-09): https://cdn.clinicaltrials.gov/large-docs/36/NCT04779736/Prot_001.pdf
  • Informed Consent Form (2024-04-05): https://cdn.clinicaltrials.gov/large-docs/36/NCT04779736/ICF_002.pdf